CLINICAL TRIAL: NCT04295850
Title: Antenatal Platelet Response On Aspirin and Correlation With HDP (Hypertensive Disorders of Pregnancy)
Acronym: APROACH
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); March of Dimes (Other)
Responsible Party: Sponsor
Other Study IDs: 19F.887; R21HD101127 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-03-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples collected prospectively prior to aspirin initiation, after aspirin initation, and in the third trimester
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Low Dose Aspirin: Pregnant singletons at high risk for preeclampsia based on:
  * at least one high risk factor for preeclampsia: prior preeclampsia, chronic hypertension, pregestational diabetes, lupus, antiphospholipid antibody syndrome, or chronic kidney disease. OR
  * at least two of the following: BMI>30, black race, state insurance, IVF pregnancy, advanced maternal age, nulliparous or >10yr from last delivery, prior adverse pregnancy outcome
  who are planning to, but have not yet started, aspirin therapy <16 weeks' gestation. Patients will take 81mg aspirin as prescribed.
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Aspirin 81mg daily PO

SUMMARY:
This proposal has three aims to characterize the relationship between aspirin therapy, platelet function response, and prevention of hypertensive disorders of pregnancy (HDP) through a prospective, cohort study using pharmacokinetics, pharmacodynamics, pharmacogenomics and bioinformatics. The results of this proposal will provide necessary data for prospective study on individualized aspirin dose adjustment for prevention of HDP.

DETAILED DESCRIPTION:
This proposal has four aims to characterize the relationship between aspirin therapy, platelet function response, and prevention of HDP through a prospective, cohort study using pharmacodynamics, pharmacogenomics and bioinformatics. The results of this proposal will provide necessary data for prospective study on individualized aspirin dose adjustment for prevention of HDP.

Aim 1: Establish pharmacodynamic endpoints for aspirin in prevention of HDP Hypothesis: PFA-100 closure time and serum thromboxane/urinary dehydrothromboxane-B2 (dTX-B2) are pharmacodynamic markers of aspirin response and are predictive of HDP high risk pregnant patients.

Aim 2: Explore aspirin pharmacogenetics by assessing the relationship between platelet receptor genotype, aspirin response, and prevention of HDP Hypothesis: Platelet receptor genotype is associated with race and may result in reduced platelet response to aspirin therapy, and increased incidence of HDP.

Aim 3: Assess the utility of circulating microRNA as a marker of aspirin response in pregnancy and risk of HDP Hypothesis: Quantitative expression of selected miRNAs are biomarkers for response to aspirin therapy and risk of HDP.

Aim 4: Evaluate aspirin pharmacokinetics/pharmacodynamics Hypothesis: Individual factors influence aspirin pharmacokinetics/pharmacodynamics and may impact individual dosing of aspirin

ELIGIBILITY:
Inclusion Criteria:

* Pregnant singleton, <16 weeks' gestation
* At least one high risk factor for preeclampsia: prior preeclampsia, chronic hypertension, pregestational diabetes, chronic kidney disease, lupus, antiphospholipid antibody syndrome

Exclusion Criteria:

* Contraindication to aspirin
* Current or planned use of any other anticoagulation
* Use of aspirin in pregnancy prior to enrollment
* Known platelet disorder at time of enrollment

Ages: 10 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pregnant patients at high risk for preeclampsia
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Aim 1: PFA-100 closure time and risk of hypertensive disorder of pregnancy (HDP) | 8 months (delivery)
  Difference in first trimester PFA-100 closure time between patients started on aspirin who do and do not develop HDP
Aim 2: Pharmacogenomics of aspirin | 2 weeks
  Difference in PFA-100 closure time with aspirin therapy based on platelet receptor genotype
Aim 3: MicroRNAs and HDP | 8 months (delivery)
  Regression analysis to evaluate how miRNAs 223, 126, 155, 181a, 18a, 16 levels in first trimester are associated with risk of HDP
Aim 4: Aspirin pharmacokinetics in pregnancy | 2 weeks
  Define population based pharmacokinetic model of aspirin in first trimester of pregnancy taking into consideration individual factors (gestational age, race, BMI, genotype)

SECONDARY OUTCOMES:
Aim 1: Aspirin response | 2 weeks
  Multiple logisitic regression analysis to evaluate factors (BMI, race, gestational age, genotype) associated with rate of nonresponse to aspirin therapy defined as (PFA-100>150s)
Aim 1: Prediction of HDP | 8 months (delivery)
  ROCC curve to determine threshold PFA-100 closure time after 1 week of aspirin therapy that is predictive of HDP
Aim 1: First trimester serum thromboxane and risk of HDP | 8 months (delivery)
  Comparison between first trimester serum thromboxane in those with and without hypertensive disorder of pregnancy
Aim 1: Third trimester serum thromboxane and risk of HDP | 8 months (delivery)
  Comparison between third trimester serum thromboxane in those with and without hypertensive disorder of pregnancy
Aim 2: Pharmacogenomics and Pregnancy outcome | 8 months (delivery)
  Multiple regression analysis taking into consideration platelet receptor genotype, race, BMI, and other clinical characteristics and prediction of HDP
Aim 3: MicroRNA profile and aspirin therapy | 2 weeks
  Paired comparison to evaluate how miRNAs 223, 126, 155, 181a, 18a, 16 levels change before and after aspirin therapy
Aim 4: Salicylic acid level and Serum Thromboxane | 2 weeks
  Association between serum salicylic acid with aspirin therapy and serum thromboxane with aspirin therapy
Predictors of preterm birth | 8 months (delivery)
  Multivariable logistic regression to evaluate markers predictive of preterm birth
Predictors of preeclampsia | 8 months (delivery)
  Multivariable logistic regression to evaluate markers predictive of preeclampsia and preterm preeclampsia

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared upon individual request after publication of planned analyses